CLINICAL TRIAL: NCT03260855
Title: Evaluation Study of Fear of Cancer Recurrence: Detection, Measure and Risk Factors in Lymphoma Survivorship
Acronym: PResEnCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/16/8823; 2017-A01208-45 (Other: ID-RCB)
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Lymphoma
Keywords: Lymphoma; Cancer survivorship; Fear
MeSH Terms: conditions — Lymphoma | interventions — Surveys and Questionnaires; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lymphoma survivorship (Other): This present study is based on an interventional (with an analysis of human blood sample) and on the use of different Questionnaires/Scales.
  Interventions: Other: Questionnaires/Scales; Other: Human blood sample

INTERVENTIONS:
Other: Questionnaires/Scales — Scale of Fear of Cancer Recurrence Inventory, Hospital Anxiety and Depression Scale, Evaluation of stress and life quality.
Other: Human blood sample — The intervention is based on blood test.

SUMMARY:
Cancer survivorship has become an important aspect of oncology research due to the risk of physical and psychosocial complications. These latter concerns 50 % of patients. So, the aim of this research is to measure frequency and intensity of one of these issues: the fear of cancer recurrence (FCR) in the lymphoma survivorship beginning, at M0.

DETAILED DESCRIPTION:
Indeed, in a recent work published by our team, several complication types in cancer survivorship has been identified: physical but also psychosocial disorders, which can lead to quality of life deterioration. The FCR in lymphoma pathology isn't yet documented and only a few studies concern the risk factors determination (age, sex, disease stage, treatment type, level of education, co-morbidity, isolation (familial status), financial resources, character trait in others cancers. Moreover, the FCR can be amplified by familial (young children) or professional responsibilities (self-employed profession). The consequences of FCR are poorly evaluated and are, however, potentially manifold: psychologic disorders, psychotropic consummation, delay of return to work and quality of life deterioration.

So, FCR is an innovating research project, which studies the FCR incidence in the beginning of lymphoma After-Cancer (AC) M0 and also the associated risk factors we can class in three types: 1. "Patient" factors (age, sex, habitat: rural/urban, familial status, level of education, financial resources, co-morbidity), 2. "disease" factors: histological type, disease stage, risk factor, 3. "treatment" factors : conventional versus intensified. Moreover, we will study the consequences of FCR M0 upon quality of life and if there is a need of psychotherapy from the very beginning of after-cancer phase, for high intensity FCR.

This present study is based on an interventional (with an analysis of human blood sample) prospective cohort, treated with anthracycline-containing regimens. This is a monocentric study which takes place in the Institut University du Cancer of Toulouse. The evaluation uses the scale of Fear of Cancer Recurrence Inventory (FCRI). The inclusion period lasts 2 years and patients will be followed during 2 years with a measure at M0, M12 and M24.

ELIGIBILITY:
Inclusion Criteria:

* Complete response of lymphoma (Cheson criteria 2007) after initial treatment
* Malin lymphoma (Hodgkin or not) treated with anthracyclines for at least 6 cycles : Adriamycin, Bleomycin, Vinblastine, and Dacarbazine (ABVD) or BEACOPP, Cyclophosphamide, hydroxydaunomycin, Oncovin, and prednisone (CHOP) et Rituximab (R-CHOP), miniCHOP et RminiCHOP, RACVBP having received or not an intensification with autologous hematopoietic stem cell transplantation in first-line
* Registered the consent to be included in this study

Exclusion Criteria:

* Person under judicial protection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2023-03-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients developing a Fear of Cancer Recurrence according to the scale of Fear of Cancer Recurrence Inventory. | Day 0, Month 12 and Month 24
  A score greater than or equal to 13 in the under-scale 2 of Fear of Cancer Recurrence Inventory (severity) represents the threshold value and a greater score than 19/32 indicates a very intensive Fear of Cancer Recurrence.

SECONDARY OUTCOMES:
Analysis of "Patient" factors | Day 0
  Patient's age, sex, accommodation, marital status, education level, resources, co-morbidity, personal story/Paykel scale, and biological stress' marker are evaluated.
Analysis of "disease" factors | Day 0
  Histologic type, disease stade and risk factors (Hasenclever score, Prognostic index for lymphoma (B or T) and Prognostic index for follicular lymphoma) are evaluated.
Analysis of "Treatment" factors | Day 0
  Conventional treatment versus intensify treatment and adverse effects (grade CTCAE ≥3) are evaluated.
Analysis of psychological disorders | Day 0, Month 12 and Month 24
  Anxiety and depression measured by Hospital Anxiety and Depression Scale and stress' evaluation.
Analysis of scale of Fear of Cancer Recurrence Inventory and life's quality association | Day 0, Month 12 and Month 24
  Life's quality is evaluated by 36-Item Short Form Survey.
Analysis of trigger factors and coping | Day 0, Month 12 and Month 24
  Score of category 1 and 4 of Fear of Cancer Recurrence Inventory are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Laurent, Pr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Institut Universitaire du Cancer de Toulouse CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barboza Solis C, Kelly-Irving M, Fantin R, Darnaudery M, Torrisani J, Lang T, Delpierre C. Adverse childhood experiences and physiological wear-and-tear in midlife: Findings from the 1958 British birth cohort. Proc Natl Acad Sci U S A. 2015 Feb 17;112(7):E738-46. doi: 10.1073/pnas.1417325112. Epub 2015 Feb 2. PMID 25646470
- [Background] Bertuccio P, Bosetti C, Malvezzi M, Levi F, Chatenoud L, Negri E, La Vecchia C. Trends in mortality from leukemia in Europe: an update to 2009 and a projection to 2012. Int J Cancer. 2013 Jan 15;132(2):427-36. doi: 10.1002/ijc.27624. Epub 2012 May 29. PMID 22553155
- [Background] Compaci G, Rueter M, Lamy S, Oberic L, Recher C, Lapeyre-Mestre M, Laurent G, Despas F. Ambulatory Medical Assistance--After Cancer (AMA-AC): A model for an early trajectory survivorship survey of lymphoma patients treated with anthracycline-based chemotherapy. BMC Cancer. 2015 Oct 24;15:781. doi: 10.1186/s12885-015-1815-7. PMID 26498342
- [Background] Koch L, Bertram H, Eberle A, Holleczek B, Schmid-Hopfner S, Waldmann A, Zeissig SR, Brenner H, Arndt V. Fear of recurrence in long-term breast cancer survivors-still an issue. Results on prevalence, determinants, and the association with quality of life and depression from the cancer survivorship--a multi-regional population-based study. Psychooncology. 2014 May;23(5):547-54. doi: 10.1002/pon.3452. Epub 2013 Nov 30. PMID 24293081
- [Background] McGinty HL, Small BJ, Laronga C, Jacobsen PB. Predictors and patterns of fear of cancer recurrence in breast cancer survivors. Health Psychol. 2016 Jan;35(1):1-9. doi: 10.1037/hea0000238. Epub 2015 Jun 1. PMID 26030308
- [Background] Mehnert A, Koch U, Sundermann C, Dinkel A. Predictors of fear of recurrence in patients one year after cancer rehabilitation: a prospective study. Acta Oncol. 2013 Aug;52(6):1102-9. doi: 10.3109/0284186X.2013.765063. Epub 2013 Feb 5. PMID 23384721
- [Background] Simard S, Savard J, Ivers H. Fear of cancer recurrence: specific profiles and nature of intrusive thoughts. J Cancer Surviv. 2010 Dec;4(4):361-71. doi: 10.1007/s11764-010-0136-8. Epub 2010 Jul 10. PMID 20617394
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Spector DJ, Noonan D, Mayer DK, Benecha H, Zimmerman S, Smith SK. Are lifestyle behavioral factors associated with health-related quality of life in long-term survivors of non-Hodgkin lymphoma? Cancer. 2015 Sep 15;121(18):3343-51. doi: 10.1002/cncr.29490. Epub 2015 Jun 2. PMID 26036473